CLINICAL TRIAL: NCT06355232
Title: A Binded, Randomised, Controlled Cross-over Trial to Assess the Safety and Efficacy of Mucosal Covid-19 and Influenza Vaccines
Brief Title: Covid-19 and Influenza Oral Vaccine Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Australian Respiratory and Sleep Medicine Institute Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Vaxine-2301
Record Dates: First submitted 2024-04-07; First posted 2024-04-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: covid19 Infection; Influenza, Human
Keywords: covid-19; influenza; pandemic; mucosal; spikogen; advax; adjuvant; vaccine
MeSH Terms: conditions — COVID-19; Influenza, Human | interventions — COVID-19 Vaccines; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Randomised, controlled cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A comparator vaccine (influenza) with an identical appearance will be used as the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Covid-19 vaccine group (Experimental): Subjects in this group will receive two sublingual doses of COVID-19 vaccine two weeks apart. Three months after the second dose they will receive two sublingual doses of influenza vaccine two weeks apart.
  Interventions: Biological: Covid-19 vaccine; Biological: Influenza vaccine
- Influenza vaccine group (Experimental): Subjects in this group will receive two sublingual doses of influenza vaccine two weeks apart. Three months after the second dose they will receive two sublingual doses of COVID-19 vaccine two weeks apart.
  Interventions: Biological: Covid-19 vaccine; Biological: Influenza vaccine
- Combined vaccine group (Experimental): Subjects in this group will receive two sublingual doses of combined COVID-19 and influenza vaccine two weeks apart. Three months after the second dose they will receive two sublingual doses of placebo vaccine two weeks apart.
  Interventions: Biological: Covid-19 vaccine; Biological: Influenza vaccine

INTERVENTIONS:
Biological: Covid-19 vaccine — Recombinant SARS-CoV-2 spike protein with Advax-CpG55.2 adjuvant
  Other Names: SARS-CoV-2 vaccine
Biological: Influenza vaccine — Inactivated seasonal influenza vaccine with Advax-CpG55.2 adjuvant

SUMMARY:
The purpose of the current study is to assess the effectiveness of protein-based COVID-19 or influenza vaccines when given individually or together via oral/ sublingual mucosal route instead of intramuscular delivery. The comparator will be a seasonal influenza vaccine which will also be administered with Advax-CpG adjuvant via the oral route. This study will use a cross-over design and everyone in the study will over a space of about 4 months receive both the COVID-19 and influenza vaccines.

DETAILED DESCRIPTION:
The SARS-CoV-2 outbreak has caused millions of deaths globally. It has a particularly high mortality rate in elderly people and those with chronic disease. SARS-COV-2 vaccines remain a key priority to help fight the current pandemic as they help reduce symptomatic infection and disease severity. However, vaccine immunity starts to wane as early as 3 months following the most recent immunisation. This rapidly waning vaccine immunity is a particular problem for the newer Omicron variants. Spikogen® vaccine is an Advax-CpG55.2 adjuvanted recombinant protein vaccine that was shown to significantly reduce infection and serious disease in a pivotal Phase 3 trial in 16,876 participants who received two intramuscular doses 3 weeks apart. SpikoGen® vaccine was licensed for use in the Middle East as a primary vaccine course in adults in October 2021. Eight million doses of SpikoGen® vaccine have subsequently been supplied to date. A booster study confirmed the safety and immunogenicity of SpikoGen® vaccine when given as a third dose intramuscular booster to adult participants who previously received two doses of either inactivated viral vaccine, adenoviral vector vaccine, mRNA or recombinant protein vaccine. While COVID-19 vaccines such as SpikoGen® vaccine have been shown to reduce the incidence of severe SARS-CoV-2 infection disease, they have less effect on SARS-CoV-2 infection or transmission. This is because intramuscular vaccines largely work by increasing antibody and T cell levels within the body, whereas what is needed to prevent infection and transmission is mucosal immunity, which means increasing immunity at the body surfaces where the virus initially gets access to the body, namely the mucosal surfaces of the nose and upper respiratory tract. To induce mucosal immunity normally requires immune cells at these respiratory tract surfaces to be exposed to the relevant viral antigen, which requires the vaccine to be applied to these surfaces in such a way as to trigger an appropriate immune response.The current study is based on the finding that an adjuvanted protein-based COVID-19 vaccine (SpikoGen®) when given as 2 sublingual doses 2 weeks apart in monkeys that had previously received a primary course of 2 intramuscular doses of the same vaccine, was safe and well tolerated and induced robust protection against challenge with the heterologous Omicron BA.5 virus. The monkeys that received the sublingual boost also showed reduced nasal virus shedding (additional details in the Investigator Brochure). This suggests an oral/ sublingual COVID-19 vaccine may also help block virus transmission. Similarly, mice that received sublingual inactivated influenza vaccine with Advax-CpG adjuvant have demonstrated robust protection against an otherwise lethal influenza infection. The purpose of the current study is to assess the effectiveness of protein-based COVID-19 or influenza vaccines when given individually or together via oral/ sublingual mucosal route instead of intramuscular delivery. The comparator will be a seasonal influenza vaccine which will also be administered with Advax-CpG adjuvant via the oral route. This study will use a cross-over design and everyone in the study will over a space of about 4 months receive both the COVID-19 and influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Males or females 18 years of age or older
* Understand and are likely to comply with planned study procedures and be available for all study visits.
* Do not plan to have a non-study COVID-19 or influenza vaccine within the next 6 months.

Exclusion Criteria:

* Allergy to COVID-19 or seasonal influenza vaccine or one of its components e.g. polysorbate 80.
* Have received a COVID-19 or influenza vaccine or an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent or a COVID-19 or influenza vaccine during the trial reporting period.
* Any serious medical, social or mental condition which, in the opinion of the investigator, would be detrimental to the subjects or the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 Seroconversion | Between baseline and 2 weeks post the second dose
  Proportion of study participants who seroconvert (4-fold or greater rise in serum spike antibody) by primary vaccine group
Influenza Seroconversion | Between baseline and 2 weeks post the second dose
  Proportion of study participants who seroconvert (4-fold or greater rise in hemagglutinin antibody) by primary vaccine group
SARS-CoV-2 Seroprotection | Between baseline and 2 weeks post the second dose
  Proportion of study participants who achieve a spike protein neutralisation titer of 32 or greater by primary vaccine group
Influenza Seroprotection | Between baseline and 2 weeks post the second dose
  Proportion of study participants who achieve a hemagglutinin neutralisation titer of 40 or greater by primary vaccine group
SARS-CoV-2 Geometric mean titer fold change | Between baseline and 2 weeks post the second dose
  Increase in Geometric mean titer of spike neutralisation antibodies by primary vaccine group
Influenza geometric mean titer fold change | Between baseline and 2 weeks post the second dose
  Increase in Geometric mean titer of spike neutralisation antibodies by primary vaccine group
Safety assessment 1 | Between time of administration of first dose and through study completion, an average of 10 months
  Frequency of Adverse events by primary vaccine group
Safety assessment 2 | Between time of administration of first dose and through study completion, an average of 10 months
  Frequency of Serious Adverse events by primary vaccine group
SARS-CoV-2 infection | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  Frequency of SARS-CoV-2 infections in study participants by primary vaccine group, age, gender, co-morbidities, and past infection
Influenza infection | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  Frequency ofinfluenza infections in study participants by primary vaccine group, age, gender, co-morbidities, and past infection

SECONDARY OUTCOMES:
Antibody durability | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  The proportion of subjects who remain seroprotected throughout the duration of the study including broken down by primary vaccine group.
Seroconversion in participants with and without evidence of past infection | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  Antibody seroconversion in participants by primary vaccine group
Antibody GMT in participants with and without evidence of past infection | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  Antibody GMT in baseline seropositive versus negative participants by primary vaccine group.
Antibody correlates of protection | From 2 weeks post the administration of the second dose and through study completion, an average of 10 months
  antibody levels in subjects with or without breakthrough infection

CONTACTS AND LOCATIONS:
Overall Officials: Dimitar Sajkov, MBBS/PhD, Principal Investigator — ARASMI
Locations (1):
- ARASMI, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with external researchers